CLINICAL TRIAL: NCT03215914
Title: Effect of Hybrid Closed-Loop Insulin Delivery on Glucose Counterregulation in Long Standing Type 1 Diabetes: A Proof of Concept, Mechanistic, Single-Arm Clinical Trial
Brief Title: Hybrid Closed Loop Insulin Delivery System in Hypoglycemia
Acronym: Aim2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael R. Rickels, MD, MS, Professor of Medicine, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 827557; 2R01DK091331 (NIH)
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Type1diabetes; Hypoglycemia Unawareness; Nocturnal Hypoglycemia; Hypoglycemia Night; Hypoglycemia
Keywords: Closed loop insulin delivery system; Insulin Pump; Glycemic control; Glucose Counterregulation
MeSH Terms: conditions — Hypoglycemia | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Open label, single-arm trial of the effect of hybrid closed-loop insulin delivery on glucose counterregulatory mechanisms assessed by the stepped- hyperinsulinemic hypoglycemic clamp in patients with long standing type 1 diabetes complicated by hypoglycemia unawareness.
Masking Description: No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects with type 1 diabetes using MiniMed 670G system (Experimental): Eligible subjects with type 1 diabetes will initiate hybrid closed-loop insulin delivery based on interstitial glucose monitoring via the MiniMed 670G system according to Medtronic's labeling. This system combines subject-delivered pre-meal boluses with automatic interprandial insulin delivery that includes automated functions for both predictive and threshold suspension of insulin delivery intended to minimize exposure to glucose levels < 70 mg/dl.
  Interventions: Device: MiniMed 670G system

INTERVENTIONS:
Device: MiniMed 670G system — Eligible subjects with type 1 diabetes will initiate hybrid closed-loop insulin delivery based on interstitial glucose monitoring via the MiniMed 670G system according to Medtronic's labeling. This system combines subject-delivered pre-meal boluses with automatic interprandial insulin delivery that includes automated functions for both predictive and threshold suspension of insulin delivery intended to minimize exposure to glucose levels < 70 mg/dl.

SUMMARY:
Can a type 1 diabetic adult avoid low glucoses and regain hypoglycemia awareness using a hybrid closed loop insulin delivery system? Involvement is 22 months (13 visits) and includes a 4-week Screening Phase and an 18-month Intervention Phase. Participants will undergo 3 Hyperinsulinemic Clamps done at: Baseline (before starting the device and after completing the screening), 6 months (after using the device 6 months), and after using the device for 18 months. This metabolic testing will allow us to measure improvement in hypoglycemia awareness.

DETAILED DESCRIPTION:
The purpose of this small, proof-of-concept, mechanistic study is to determine whether hybrid closed-loop insulin delivery can achieve sufficient hypoglycemia avoidance in patients with long standing type 1 diabetes experiencing hypoglycemia and symptom unawareness despite receiving intensive insulin therapy standard-of-care to improve glucose counterregulation against insulin-induced hypoglycemia. As it remains critically important to understand the potential physiologic benefits of hypoglycemia avoidance by means of a hybrid closed-loop system in this population, studying each well characterized subject as his/her own control by a within subject design should serve the study purpose, and has been the standard approach to assessing the effects of various approaches to hypoglycemia avoidance in patients with unawareness. The data generated will be available to power future randomized clinical trials to determine the comparative efficacy of emerging artificial pancreas and β-cell replacement approaches to achieve target glycemic control with amelioration of problematic hypoglycemia in type 1 diabetes.

Screening Phase At the screening visit, the study details and procedures will be discussed with a research coordinator and at least one of the PI or the research nurse practitioner. The potential participant is given adequate time to ask questions and review the informed consent document. Once satisfied that all questions have been answered, the potential participant will either decline to participate or sign the informed consent document. This may occur at a subsequent visit if the potential participant desires, in order to think further about what participation means and/or to consult with family, friends and/or a personal physician. The consent form is signed in the presence of a witness (research coordinator +/- family member). All participants must read, sign, and date a consent form before entering the study, undergoing physical examination or undergoing any testing. The informed consent form will be revised whenever important new safety information is available, whenever the protocol is amended, and/or whenever any new information becomes available that may affect participation in the studies.Eligibility will be confirmed through the performance of a history and physical examination by the PI or the research nurse practitioner, EKG, urine pregnancy test (if applicable), serum chemistries, TSH, cell counts, HbA1c and C-peptide, completion of glycemic lability and hypoglycemia awareness and hypoglycemia severity questionnaires, placement of a 7 day blinded CGM (iPro 2, Medtronic Diabetes, Northridge, CA) unless on CGM available for downloading, and 7 day accelerometry (WGT3X-BT, Actigraph LLC,) to define the nocturnal period.

Only after all eligibility criteria (inclusion and exclusion) are met, will a potential subject be enrolled. Repeated clinical testing throughout the study will ensure the continued safety and minimization of risk for the enrolled participants.

Study Intervention Phase Eligible subjects will complete a baseline assessment of glucose counterregulation by stepped- hyperinsulinemic hypoglycemic clamp prior to starting intervention with the hybrid closed-loop system (MiniMed 670G system, Medtronic Diabetes, Northridge, CA). Unless this system becomes available to the subject via their insurance carrier, one will be provided for them. Subjects will also receive a study glucometer (Contour Next Link 2.4, Bayer, Indianapolis, IN) that communicates with the MiniMed 670G insulin pump for bolus dosing calculation and glucose sensor calibration. Subjects who cannot maintain > 80% (or 6/7 day) compliance with the sensor component as assessed at each study visit may be dropped since less compliance has not been associated with any benefit of CGM to glycemic control and limits the potential for benefit from LGS on hypoglycemia avoidance. Accuracy of the sensor will be assessed at each visit through devise download and interpretation. Study visits will occur weekly for the first month, then monthly until month 6, and then every 3 months until month 18. This schedule will allow for determination of possible benefit from hybrid closed- loop insulin delivery on glucose counterregulation after 6 months of intensive provider support, and then for assessment of the durability or potential further gains in beneficial effects after another 12 months of more typical provider interaction occurring every 3 months. Weekly visits may be performed via telephone with uploading devise data to Care Link for review and interpretation. Uploaded or downloaded insulin delivery, blood and sensor glucose monitoring, insulin dose settings and CGM calibration accuracy, alert settings, time spent in auto and manual modes, and LGS threshold and activity will be assessed at each visit, targeting > 80% CGM and LGS compliance, adjusting basal and bolus insulin dosing in order to minimize glycemic excursions while maximizing hypoglycemia (< 60 mg/dl) avoidance, with adjustment of alarms set to alert the subject to rapidly increasing or decreasing glucose and predict the occurrence of elevated or low blood glucose. During manual mode, target glucose ranges will be 90 - 140 mg/dl before meals, < 180 mg/dl after meals, and 120 - 160 mg/dl at bedtime, with correction dosing to no lower than 100 mg/dl during the day, and 120 mg/dl overnight. Alarm settings may be individualized to target these ranges, but the hypoglycemia alarm for LGS will not be set lower than 70 mg/dl. During auto mode, the automated interprandial basal insulin delivery will adjust according to the closed-loop algorithm to target a sensor glucose of 120 mg/dl, which may be temporality increased to 150 mg/dl if needed to further minimize exposure to hypoglycemia during exercise or overnight. Prior to each 3 monthly visit, subjects will wear an actigraph monitor ( WGT3X-BT, Actigraph LLC,) for three weeks in order to define the nocturnal period. Every 6 months measures of hypoglycemia awareness (Clarke score) and severity (HYPO score), and the glycemic lability index (LI) will be calculated from questionnaires, event diaries, and device downloads, respectively. At 6 months and at 18 months, subjects will again undergo assessment of glucose counterregulation by stepped-hyperinsulinemic hypoglycemic clamp testing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 25 to 70 years.
* Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol.
* Clinical history compatible with type 1 diabetes with disease onset < 40 years of age and insulin dependent for > 10 years.
* Absent C-peptide (< 0.3 ng/ml).
* Involvement in intensive diabetes management defined as the use of basal-bolus insulin analog delivery by multi-dose injection (MDI) or continuous subcutaneous insulin infusion (CSII) together with self-monitoring of blood glucose values more than 3 times daily with or without continuous glucose monitoring (CGM) under the direction of an endocrinologist, diabetologist, or diabetes nurse practitioner with at least 3 clinical evaluations during the previous 12 months.
* Hypoglycemia unawareness manifested by a Clarke score of 4 or more AND at least 1 of the following: HYPO score greater than or equal to the 90th percentile (1047); OR marked glycemic lability defined by a glycemic lability index (LI) score greater than or equal to the 90th percentile (433 mmol/l2/h•wk-1); OR a composite of a HYPO score greater than or equal to the 75th percentile (423) and a LI greater than or equal to the 75th percentile (329) (Senior et al., 2015).
* Documented > 5% time spent in the hypoglycemic range (glucose < 60 mg/dl) by 7 day real- time or blinded CGM; at least one episode of hypoglycemic during the 7 days must occur overnight.

Exclusion Criteria:

* BMI ≥ 30 kg/m2.
* Insulin requirement of ≥ 1.0 units/kg•day.
* HbA1c ≥ 10%.
* Untreated proliferative diabetic retinopathy.
* Uncontrolled hypertension: systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
* Active cardiovascular disease
* Abnormal kidney function: eGFR < 60 ml/min/1.73 m2.
* Abnormal liver function: persistent elevation of liver function tests > 1.5 times the upper limit of normal.
* Untreated hypothyroidism, Addison's disease, or Celiac disease.
* Anemia: baseline hemoglobin concentration < 11 g/dl in women and < 12 g/dl in men.
* Presence of a seizure disorder not related to prior severe hypoglycemia.
* Use of glucocorticoids greater than 5 mg of prednisone daily, or an equivalent physiologic dose of hydrocortisone.
* For female participants of child-bearing potential: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of study participation. Oral contraceptives, intra-uterine devices, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment.
* Use of any investigational agents within 4 weeks of enrollment.
* Any medical condition that, in the opinion of the PI, will interfere with the safe completion of the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Rickels, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Clinical and Translational Research Center, Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Rodebaugh Diabetes Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania - Institute for Diabetes, Obesity and Metabolism, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
It is not yet known if there will be any further plan to make IPD available besides the Informed Consent.
Supporting Information: ICF
Time Frame: Immediately
Access Criteria: To request an informed consent document please contact:
  Ginger Bakes, CCRC: Cornelia.dalton-bakes@uphs.upenn.edu

REFERENCES:
- [Derived] Malone SK, Matus AM, Flatt AJ, Peleckis AJ, Grunin L, Yu G, Jang S, Weimer J, Lee I, Rickels MR, Goel N. Prolonged Use of an Automated Insulin Delivery System Improves Sleep in Long-Standing Type 1 Diabetes Complicated by Impaired Awareness of Hypoglycemia. J Diabetes Sci Technol. 2024 Nov;18(6):1416-1423. doi: 10.1177/19322968231182406. Epub 2023 Jul 14. PMID 37449426
- [Derived] Malone SK, Peleckis AJ, Grunin L, Yu G, Jang S, Weimer J, Lee I, Rickels MR, Goel N. Characterizing Glycemic Control and Sleep in Adults with Long-Standing Type 1 Diabetes and Hypoglycemia Unawareness Initiating Hybrid Closed Loop Insulin Delivery. J Diabetes Res. 2021 Feb 12;2021:6611064. doi: 10.1155/2021/6611064. eCollection 2021. PMID 33628834
- See also: Institute for Diabetes, Obesity and Metabolism Research Studies — https://www.med.upenn.edu/idom/trials.html
- See also: Research Studies at the University of Pennsylvania — https://clinicalresearch.itmat.upenn.edu
- See also: Perelman School of Medicine / Faculty Search / Michael Rickels, M.D., M.S — https://www.med.upenn.edu/apps/faculty/index.php/g363/c644/p32032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects With Type 1 Diabetes Using MiniMed 670G System
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 18 participants were consented. Of the 18, 6 did not meet inclusion and 2 were dropped.10 were enrolled and completed the study.
Arm/Group | Subjects With Type 1 Diabetes Using MiniMed 670G System
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Endogenous Glucose Produciton [Mean (Standard Deviation); unit: [mg/(kgxmin)]] | .73 (.23)

OUTCOME MEASURES:

1. Primary Outcome: Endogenous Glucose Production
Description: The primary outcome measure will be endogenous glucose production in response to insulin-induced hypoglycemia.
Time Frame: After 6 months of hybrid closed-loop insulin delivery.
Measure: Mean (Standard Deviation); unit: [mg/(kgxmin)]
Arm/Group | Subjects With Type 1 Diabetes Using MiniMed 670G System
Number analyzed (Participants) | 10
[mg/(kgxmin)] | .66 (.13)

2. Secondary Outcome: Endogenous Glucose Production
Description: The secondary outcome measure will be endogenous glucose production in response to insulin-induced hypoglycemia.
Time Frame: After 18 months of hybrid closed-loop insulin delivery.
Measure: Mean (Standard Deviation); unit: [mg/(kgxmin)]
Arm/Group | Subjects With Type 1 Diabetes Using MiniMed 670G System
Number analyzed (Participants) | 10
[mg/(kgxmin)] | .69 (.11)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Subjects With Type 1 Diabetes Using MiniMed 670G System
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Type 1 Diabetes Using MiniMed 670G System (N=10)
Hypoglycemia (Endocrine disorders) | 4 (5) — Hypoglycemia <54mg/dL requiring 3rd party assistance
URI (Infections and infestations) | 2 (2)
Bacterial Infections (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03215914/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT03215914/ICF_001.pdf